CLINICAL TRIAL: NCT02687009
Title: A Phase I Study of Niclosamide in Patients With Resectable Colon Cancer
Brief Title: A Study of Niclosamide in Patients With Resectable Colon Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Michael Morse, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Morse, MD, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00066964
Record Dates: First submitted 2016-02-10; First posted 2016-02-22 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Colon Cancer
Keywords: colon cancer; Wnt pathway; Frizzled
MeSH Terms: conditions — Colonic Neoplasms | interventions — Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niclosamide (Experimental)
  Interventions: Drug: Niclosamide

INTERVENTIONS:
Drug: Niclosamide — Niclosamide will be taken orally in the morning of each day from day 1-7 prior to surgery for resection of primary tumor. Niclosamide tablets must be chewed well prior to swallowing.
  Other Names: Yomensan

SUMMARY:
This study evaluates the safety of Niclosamide in patients with colon cancer that are undergoing primary resection of their tumor. This is a phase I study with three dosage levels to determine the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
Niclosamide is a drug traditionally used in parasitic infections that has recently been shown to regulated the Wnt signaling pathway in cells at the level of the Frizzled receptor.

The Wnt pathway is critical for embryogenesis, differentiation of progenitor cells, and supports proliferation of neoplastic tissue. In cancer, activation of the Wnt pathway leads to increased transcription of genes important for growth, proliferation, differentiation, apoptosis, genetic stability, migration, and angiogenesis. The Wnt pathway has particular importance in colorectal cancer.

The purpose of this study is to obtain safety data along with pharmacokinetic data and information on the changes in the WNT pathway signalling following niclosamide administration in humans. This phase I study will support future studies in patients with more advanced cancer and other cancers with dysregulation of the Wnt pathway.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colon adenocarcinoma with a plan to undergo surgical resection no sooner than 7 days from the projected date of study drug initiation. Patients with rectal cancer not receiving pre-operative chemoradiotherapy are also eligible.
* Karnofsky performance status greater than or equal to 70%
* Age ≥ 18 years.
* Adequate hematologic function, with ANC > 1500/microliter, hemoglobin ≥ 9 g/dL (may transfuse or use erythropoietin to achieve this level), platelets ≥ 100,000/microliter; INR <1.5, PTT <1.5X ULN
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board's guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up, as required by this protocol.

Exclusion Criteria:

* Patients with concurrent cytotoxic chemotherapy or radiation therapy are excluded
* Known active brain or leptomeningeal metastases (defined as symptomatic metastases) or continued requirement for glucocorticoids for brain or leptomeningeal metastases. Treated, asymptomatic metastases are permitted provided the patient has been off steroids for at least 1 month prior to day 1 of study drug.
* Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
* Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
* Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other carcinoma in situ that has been treated.
* Presence of a known active acute or chronic infection including: a urinary tract infection, HIV or viral hepatitis.
* Patients with prior use of niclosamide or allergies to niclosamide will be excluded from the protocol.
* Concomitant use of strong CYP3A4, CYP 1A2 , or CYP2C9 substrates (See http://medicine.iupui.edu/clinpharm/ddis/main-table).
* Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 12 months following the last dose of niclosamide. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
* Patients with complete bowel obstruction or who are at high risk for GI perforation or severe hemorrhage. Patients with inflammatory bowel disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 5 DAYS
  The NCI Common Toxicity Criteria version 4.0 will be used to grade adverse events to determine dose limiting toxicity for safety measure
Dose limiting toxicity | 30 DAYS
  he NCI Common Toxicity Criteria version 4.0 will be used to grade adverse events to determine dose limiting toxicity for safety measure

SECONDARY OUTCOMES:
Niclosamide blood levels | 1 DAY
Niclosamide blood levels | 2 days
Niclosamide blood levels | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osada T, Chen M, Yang XY, Spasojevic I, Vandeusen JB, Hsu D, Clary BM, Clay TM, Chen W, Morse MA, Lyerly HK. Antihelminth compound niclosamide downregulates Wnt signaling and elicits antitumor responses in tumors with activating APC mutations. Cancer Res. 2011 Jun 15;71(12):4172-82. doi: 10.1158/0008-5472.CAN-10-3978. Epub 2011 Apr 29. PMID 21531761